CLINICAL TRIAL: NCT00893178
Title: Impact of Different Genetic Polymorphism on the Pulmonary Pressure in Patients With Pulmonary Hypertension of Different Cause With Special Focus on Patients With Chronic Heart Failure
Brief Title: Impact of Polymorphism on Pulmonary Pressure in Subjects With Pulmonary Hypertension of Different Cause
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, PI, University of Leipzig
Other Study IDs: SMW 03
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Congestive Heart Failure; Pulmonary Hypertension
Keywords: eNOS Polymorphism; TNF alpha polymorphism; pulmonary pressure; polymorphism of vasoactive substances
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA Blood, Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CHF with elevated PAP: CHF patients (LVEF > 35%) with elevated mean pulmonary pressure( > 20 mmHg ) measured by pa catheter
- CHF patient without elevated PAP: CHF patients (LVEF > 35%) with normal mean pulmonary pressure
- Normal EF with elevated PAP: Patients with normal LVEF < 60% with elevated mean pulmonary pressure

SUMMARY:
Pulmonary Hypertension (PH) is a disease that is characterized by vasoconstriction of small vessels of the lung. Many cases do have proliferation of endothelial cells within these vessels. A possible influence of polymorphisms of genes relevant for inflammatory and endothelial processes is suspected.

Especially patients with chronic heart failure can develope PH. The reasons therefore are lacking.

The researchers investigate different polymorphism and the influence of these on pulmonary artery pressure (measured invasively) in patients with congestive heart failure (CHF) and patients with primary pulmonary hypertension.

DETAILED DESCRIPTION:
The study consists of 3 arms-patients with CHF and PH, patients with CHF without PH and patients without CHF and PH.

The PH measurement is due to routine catheterization, thereafter we measure different vasoactive polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* CHF with or without pulmonary hypertension or
* patients with normal LVEF and pulmonary hypertension
* right heart catheterization due to routine
* informed consent

Exclusion Criteria:

* no right heart catheterization
* no informed consent
* elevated pulmonary pressure due to valve diseases or congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHF elevated pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Correlation of the Expression of Glu 298ASP Polymorphism with pulmonary pressure | Dec. 2010

SECONDARY OUTCOMES:
Rate of G308A TNF alpha polymorphism within the different groups | Dec. 2010

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, M.D, Principal Investigator — University Leipzig-Heart Center
Locations (1):
- Heart Center Leipzig- University Leipzig, Leipzig, Germany